CLINICAL TRIAL: NCT02180607
Title: Neuronal Responses to Social Feedback in Major Depressive Disorder
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, David Hsu, Research Assistant Professor, University of Michigan
Other Study IDs: K01MH085035 (NIH)
Record Dates: First submitted 2014-06-30; First posted 2014-07-02 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Major Depressive Disorder
Keywords: depression; social; rejection; acceptance; fMRI; reward; exclusion
MeSH Terms: conditions — Depressive Disorder, Major; Depression; Rejection, Psychology

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — saliva
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Healthy Controls: Response to social feedback, monetary incentive delay, and go/no-go tasks
- MDD patients: Response to social feedback, monetary incentive delay, and go/no-go tasks

SUMMARY:
The overall goal of the proposed project is to investigate the neuronal pathways regulating the effects of social acceptance and rejection in healthy controls and patients with Major Depressive Disorder (MDD). Social acceptance and rejection are defined as the explicit declaration that an individual is liked or not liked. Social acceptance can boost one's self-esteem and mood, whereas rejection can lower them. The neurological relationship between social acceptance/rejection and depressive symptoms is not known. Using functional magnetic resonance imaging (fMRI), it is hypothesized that social feedback will activate a specific interconnected neuronal pathway involved in social separation and reward. Executive functioning and response to monetary reward will also be assessed during fMRI using two additional tasks (monetary incentive delay, parametric go no-go) to determine how these cognitive brain functions regulate responses to social feedback.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between 18 and 55 years of age
* No use of psychotropic medications in the past 4 weeks
* No regular tobacco use, and who are able to make decisions for his or her self -Patients who meet criteria for (DSM-IV) Major Depressive Disorder or Depressive Disorder Not Otherwise Specified, with Hamilton Depression Rating Scale scores ≥ 10, and may be on monotherapy (treatment for MDD with a single SSRI)
* MDD patients will be matched with healthy controls for age and education.

Exclusion Criteria:

* No serious medical illnesses or major physiological disturbance during the past three months (e.g., serious infections or pregnancy) or anemia Any other Axis I psychiatric disorder
* Pharmacological exclusion criteria include the use of psychoactive substances during past 3 months (e.g., barbiturates, anticonvulsants glutethimide, alpha-methyl dopa, corticosteroids [oral or topical creams], opiates or codeine, cyproheptadine, opioid analgesics, antipsychotic drugs)
* History of DSM-IV alcohol or drug dependence within the past 5 years
* Drug or alcohol abuse in the past 2 years or a CAGE Alcohol Screening Inventory score of >3
* Regular alcohol use during the past 6 months equal to or greater than 16 cans of beer per week or equivalent; use of street drugs during the past 2 years
* Regular tobacco use, since nicotine stimulates cortisol secretion even in smokers;
* Major chronobiological disruption or phase shift during the preceding month (e.g., total sleep deprivation, reversal of sleep-wake cycles or trans-meridian travel)
* Childbirth or miscarriage within 6 months
* Breastfeeding within 6 months of recruitment
* Progestin-only birth controls (e.g., Cerazette, Ovrette)
* No contraindications to MRI scan including neurostimulators, metal in the body, weight over 250 pounds, and girth size incompatible for MRI scanner bore
* No non-right-handed subjects
* For healthy controls, subjects will have no history of psychiatric problems in themselves or any first-degree relatives

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Individuals diagnosed with major depressive disorder (MDD), and healthy controls
Sampling Method: Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2013-10; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
fMRI blood-oxygen-level-dependent (BOLD) response | within 30 days of informed consent
  This study will compare brain activation in healthy and depressed individuals in response to social feedback, monetary reward, and behavioral inhibition. Primary regions of interest include: the amygdala, anterior insular cortex, and the nucleus accumbens. All structures will be examined bilaterally. Arbitrary units for fMRI BOLD are used to compare activation during one condition (e.g., neutral, baseline) vs. another condition (e.g., positive social feedback, monetary reward).

CONTACTS AND LOCATIONS:
Overall Officials: David T Hsu, Ph.D., Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States